CLINICAL TRIAL: NCT07380191
Title: EFFECT OF PLAZEPOD VERSUS ELECTRICAL STIMULATION ON RISK OF FALLING IN HEMODIALYSIS PATIENTS
Acronym: HD Fall Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samia Wagdy El Said Diab, EFFECT OF PLAZEPOD VERSUS ELECTRICAL STIMULATION ON RISK OF FALLING IN HEMODIALYSIS PATIENTS, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CairoU physical therapy
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Fall Risk, Fall Prevention

STUDY DESIGN:
Intervention Model Description: Application two Devices of PlazePod Device and Electrical Stimulation for 60 patients each group 30 for 3months for 40-50age Additionally life style education program, such as: Renal nutrition Fluid control Safe physical activity Sleep hygiene, energy and managing fatigue Adherence and awareness For 3 months, there was one session every week, lasting 30 minutes and comparison between two groups
Who Masked: Participant
Masking Description: Application of PlazePod Device and Electrical Stimulation for 60 patients each group 30 for 3months for 40-50age Additionally life style education program, such as: Renal nutrition Fluid control Safe physical activity Sleep hygiene, energy and managing fatigue Adherence and awareness For 3 months, there was one session every week, lasting 30 minutes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BlazePod Training plus Lifestyle Education (Experimental): Participants in this arm will receive an interactive sensorimotor training program using the BlazePod system combined with a structured lifestyle education program. BlazePod training will focus on improving balance, reaction time, coordination, and functional mobility through static and dynamic balance tasks, reactive stepping, and lower-limb coordination exercises. Training sessions will be conducted three times per week for 30 minutes over a period of 12 weeks under the supervision of a physical therapist. In addition, participants will attend a weekly lifestyle education session addressing renal nutrition, fluid management, safe physical activity, fall prevention strategies, sleep hygiene, fatigue management, and medication adherence.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES)
- Tens plus Lifestyle Education (Active Comparator): Participants in this arm will receive neuromuscular electrical stimulation (NMES) applied to the lower limb muscles, including bilateral quadriceps and hamstrings, combined with the same structured lifestyle education program as the experimental group. NMES will be delivered using a portable electrical stimulation device with parameters adjusted to produce visible and comfortable muscle contractions. Sessions will be conducted three times per week for 30 minutes over 12 weeks under physical therapist supervision. Lifestyle education sessions will be provided once weekly and will include renal nutrition, fluid control, safe physical activity, fall prevention strategies, sleep hygiene, fatigue management, and medication adherence.
  Interventions: Device: Device + Behavioral; Device: Neuromuscular Electrical Stimulation (NMES)

INTERVENTIONS:
Device: Device + Behavioral — This intervention consists of interactive sensorimotor training using the BlazePod system, a visual stimulus-based device designed to improve balance, coordination, reaction time, and functional mobility. Participants will perform static and dynamic balance exercises, reactive stepping drills, lower-limb coordination tasks, and dual-task activities in response to visual cues emitted by the BlazePod sensors. Training sessions will be conducted three times per week, with each session lasting 30 minutes, over a total duration of 12 weeks. All sessions will be supervised by a licensed physical therapist to ensure safety and appropriate progression of exercise difficulty. The intervention aims to reduce fall risk by enhancing neuromuscular control and postural stability in hemodialysis patients.
  Arms: Tens plus Lifestyle Education
Device: Neuromuscular Electrical Stimulation (NMES) — This intervention involves the application of neuromuscular electrical stimulation to the lower limb muscles, specifically the bilateral quadriceps and hamstrings, using a portable electrical stimulation device. Surface electrodes will be placed over the motor points to elicit visible and comfortable muscle contractions. Stimulation parameters will include a frequency of 35-50 Hz, pulse width of 200-400 microseconds, and a duty cycle of 10 seconds on and 30 seconds off. Sessions will be administered three times per week for 30 minutes over 12 weeks under the supervision of a physical therapist. The intervention aims to improve muscle strength, balance, functional mobility, and reduce fall risk in hemodialysis patients.

SUMMARY:
Renal nutrition Fluid control Safe physical activity Sleep hygiene, energy and managing fatigue Adherence and awareness

DETAILED DESCRIPTION:
Application of PlazePod Device and Electrical Stimulation and comparison between them to decrease fall Risk in Hemodialysis Patients

ELIGIBILITY:
Inclusion Criteria:

* :
* Male patients aged 40 to 50 years.
* Diagnosed with end-stage renal disease and receiving maintenance hemodialysis for at least 6 months.
* Medically stable and cleared by a nephrologist to participate in physical activity and/or electrical stimulation.
* Able to ambulate independently or with minimal assistance.
* Cognitively able to understand study procedures.
* Not participating in any other structured exercise program.

Exclusion Criteria:

* Severe neurological or orthopedic disorders affecting mobility.
* Unstable cardiovascular conditions.
* Cognitive impairment or sensory deficits.
* Contraindications to neuromuscular electrical stimulation.

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-21 (Estimated); Primary Completion 2026-12-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Risk of Falling Assessed by Timed Up and Go Test (TUG) | Baseline and after 12 weeks of intervention
  Change in risk of falling measured using the Timed Up and Go (TUG) test, recorded in seconds. Lower scores indicate better functional mobility and reduced fall risk.
Balance Performance Assessed by Berg Balance Scale (BBS) | Baseline and after 12 weeks
  Change in static and dynamic balance measured using the Berg Balance Scale (BBS), scored from 0 to 56 points, with higher scores indicating better balance performance.
Lower Limb Muscle Strength | Baseline and after 12 weeks
  Change in lower limb muscle strength measured using a hand-held dynamometer, recorded in kilograms (kg).

SECONDARY OUTCOMES:
Physical Activity Level | Baseline and after 12 weeks
  Change in physical activity level measured using the International Physical Activity Questionnaire - Short Form (IPAQ-SF), expressed in MET-minutes/week.
Kidney Disease-Related Quality of Life | Baseline and after 12 weeks
  Change in quality of life measured using the Kidney Disease Quality of Life Short Form questionnaire (KDQOL-36), reported as total score.

OTHER OUTCOMES:
Adherence to Intervention Program | Throughout the 12-week intervention period
  Participant adherence to the prescribed physical intervention and lifestyle education sessions, expressed as percentage of attended sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta, Tanta, Alquarbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
"At this time, we have not decided whether individual participant data will be shared. This is due to considerations of patient privacy, confidentiality, and ongoing analysis. A decision regarding data sharing will be made after study completion and in accordance with ethical guidelines."

REFERENCES:
- See also: This website provides scientific articles and studies related to lifestyle interventions, physical exercise, and fall risk in hemodialysis patients. — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Study Protocol: LifestyleStudy2026 — https://pubmed.ncbi.nlm.nih.gov/?term=hemodialysis+fall+risk+exercise — Study protocol available for review. Additional data can be shared upon request following ethical approval.